CLINICAL TRIAL: NCT04021069
Title: Using Clinicopathomic Markers to Predict Neoadjuvant Chemotherapy Response in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. William Tran, Radiation Therapist Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 270-2018
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Invasive Ductal Breast Carcinoma; Invasive Lobular Breast Carcinoma
Keywords: radiomics; pathomics; breast cancer; machine learning; biomarkers
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Fixed tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Radiomic, pathomic, and clinical markers — This is a non-interventional study.

SUMMARY:
This study examines retrospective clinical data on patients diagnosed with breast cancer and monitor their response to neoadjuvant chemotherapy, incidence of locoregional recurrence, distant metastasis, and disease-free survival. The hypothesis of this study is that breast cancer patients who achieve a pathological complete response (pCR) to neoadjuvant chemotherapy demonstrate distinct clinicopathomic biomarker signatures.

DETAILED DESCRIPTION:
The specific aims of the study are to (1) to identify clinicopathomic biomarkers from pre-treatment core biopsies that are predictive of response to neoadjuvant chemotherapy, (2) determine patterns of metastasis from primary breast cancer to other distant sites, (3) determine the rates of local recurrence in breast cancer patients, and (4) to determine if there are significant radiomic, pathomic, and clinical markers for recurrence and distant metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be men and women age 18+
* Biopsy-confirmed diagnosis of invasive breast cancer; (ER+/-, PR+/-, HER2+/-)
* Any state of disease as described by AJCC v7 criteria
* Participants must have received and completed neoadjuvant chemotherapy

Exclusion Criteria:

* Participants who had other primary cancers prior to breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll women and men with a pathologically-confirmed diagnosis of invasive breast cancer of any stage, according to the AJCC v7 criteria.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | Up to 60 months
  Evaluating the degree of absence of residual cancer cells

SECONDARY OUTCOMES:
Time to local breast recurrence | Up to 60 months
  Evaluating the time until a recurrence event has occurred in the breast
Time to distant metastasis (months) | Up to 60 months
  Evaluating onset of distant metastasis
Time to death | Up to 60 months
  Evaluating time to cancer-related death

CONTACTS AND LOCATIONS:
Overall Officials: William T. Tran, MRT(T), PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Kasia Jerzak, M.Sc., MD, Principal Investigator — Sunnybrook Health Sciences Centre; Fang-I Lu, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymized. Digital pathology images and anonymized clinical data will be deposited into the National Cancer Institute (NCI) data sharing repository, including The Cancer Imaging Archive (TCIA). Digital pathology images will also be annotated to facilitate analysis for other investigators. Computational methods, source-codes and instructions will be deposited to the open-source coding repository, GitHub (www.github.com).
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Digital pathology images, anonymized clinical data, source codes, and computational methods will be deposited to open-source repositories.